CLINICAL TRIAL: NCT01883024
Title: Prospective Study, Insulin Pump-RT Advisor (IPRA©): a Decision Support Software for Diabetic Patients Treated by Insulin Pump and Using Continuous Glucose Monitoring. Experimental Study. Evaluation by an Expert Patient Panel.
Brief Title: Insulin Pump-RT Advisor (IPRA©): a Decision Support Software for Diabetic Patients Treated by Insulin Pump and Using Continuous Glucose Monitoring. Experimental Study. Evaluation by an Expert Patient Panel.
Acronym: IPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A00495-40; LOC 1308 (Other: Rennes University Hospital)
Record Dates: First submitted 2013-06-14; First posted 2013-06-21 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
Keywords: Real time continuous glucose monitoring, decision support software, smartphone application.
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Infusion Systems; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Type 1 diabetes (Other)
  Interventions: Other: A decision support software; Other: Insulin Pump; Other: Continuous glucose monitoring

INTERVENTIONS:
Other: A decision support software
Other: Insulin Pump
Other: Continuous glucose monitoring

SUMMARY:
The purpose of the study is to assess the relevance of the advices provided by the IPRA© smartphone application for guiding the responses of insulin pump treated type 1 diabetes patients using real-time continuous glucose monitoring.

DETAILED DESCRIPTION:
Patients will be asked to evaluate the IPRA advices by connecting to IPRA© application by using their smartphone, 30 times a week for two weeks. At the end of this two week period, a satisfaction questionnaire will be completed.

ELIGIBILITY:
Inclusion Criteria:

* men and women ≥ 18 years of age,
* patients with type 1 diabetes for more than 2 years,
* patients treated by insulin pump for more than 6 months,
* patients using of real-time continuous glucose monitoring for more than 3 months,
* patients able to evaluate the IPRA advices by connecting to IPRA© application 30 times a week,
* patient able to provide written informed consent,
* patient able to provide written non-disclosure agreement

Exclusion Criteria:

* pregnancy or breastfeeding,
* current infectious disease,
* patients with no smartphone® or Internet access,
* adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Patient agreement with the IPRA© advices: global rate of agreement, according to advice subtypes, according to blood glucose levels, according to the situations (pre or post-meal, bedtime) | 3 months
  Assessment of the relevance of the advices provided by the IPRA© smartphone application for guiding the responses of insulin pump treated type 1 diabetes patients using real-time continuous glucose monitoring.

SECONDARY OUTCOMES:
Assessment of similarity between patient decisions and IPRA© advices | 3 months
  Assessment of patient satisfaction about using IPRA© and their frequency of use.
  Recording of the changes proposed by the expert patients.
Assessment of changes proposed by the experts | 3 months
Assessment of frequency of software use | 3 months
Assessment of patient satisfaction | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Guilhem, Principal Investigator — Rennes University Hospital
Locations (1):
- Service d'Endocrinologie-Diabétologie - CHU de Rennes - Hôpital Sud, Rennes, France

REFERENCES:
- [Result] Esvant A, Lefebvre MA, Campillo-Gimenez B, Lannes M, Delamarre D, Guilhem I, Poirier JY. A Mobile Application Guiding Patients With Type 1 Diabetes Using Sensor-Augmented Insulin Pump Therapy. J Diabetes Sci Technol. 2016 Jun 28;10(4):985-6. doi: 10.1177/1932296816633486. Print 2016 Jul. No abstract available. PMID 26902791